CLINICAL TRIAL: NCT07292428
Title: An Integrated and Multi-perspective Approach to Cognitive-motor Technology Rehabilitation and Telemedicine in Frail Individuals
Brief Title: Cognitive-motor Technology Rehabilitation in Frail Individuals
Acronym: FIT4COG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7943
Record Dates: First submitted 2025-12-01; First posted 2025-12-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Frail; Sensorimotor Deficits
Keywords: Frailty; Sensorimotor impairment; Technology rehabilitation; Dual-task condition
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technological Group (G-Tec) (Experimental): G-Tec patients will undergo outpatient technological rehabilitation treatment for 4 weeks using hunova® and Senso robots, followed by home-based technological rehabilitation treatment for another 4 weeks using a tablet with cognitive exercises developed specifically for home cognitive treatment, followed by 8 weeks of observation.
  Interventions: Device: Technological rehabilitation with robotic platfom and home telerehabilitation device
- Conventional Group (G-Con) (Active Comparator): G-Con patients will undergo conventional outpatient rehabilitation treatment for 4 weeks, followed by conventional home-based rehabilitation treatment, mainly cognitive in nature, for another 4 weeks, and then 8 weeks of observation.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: Technological rehabilitation with robotic platfom and home telerehabilitation device — Technological outpatient and home rehabilitation
  Arms: Technological Group (G-Tec)
Other: Conventional rehabilitation — Conventional outpatient and home rehabilitation
  Arms: Conventional Group (G-Con)

SUMMARY:
Dual performance, which involves the simultaneous execution of motor and cognitive tasks, is a fundamental aspect of everyday functioning. In the elderly population, for example, the ability to manage dual tasks can be significantly impaired, resulting in an increased risk of falls and further cognitive decline. The ability to perform two tasks simultaneously (one motor and one cognitive) is often impaired in patients with chronic sensorimotor and/or cognitive disabilities, with repercussions on both physical and cognitive abilities. Patients with chronic sensorimotor and/or cognitive disabilities consistently show greater deficits in dual performance than healthy individuals, with repercussions on both motor and cognitive functioning. These deficits are influenced by psychological, neural, and disease-specific factors, but targeted interventions and dual-task training can help improve outcomes.

Some authors have pointed out that dual-task training can improve attention, functional mobility, and overall cognitive function more effectively than single-task training. One of the main advantages of dual-task training is the reduction of the risk of falls in the elderly population and in chronic patients with sensorimotor disorders: dual-task training has been shown to improve dynamic balance and stability, even during walking, and cognitive function.

Telerehabilitation is a branch of telemedicine that uses different types of technology to provide remote rehabilitation services. Telerehabilitation, like telemedicine, can be delivered through three distinct mechanisms: synchronous mode, in which the patient and physician communicate in real time using technological tools; remote monitoring mode, in which the patient's condition is monitored remotely; and asynchronous mode, in which there is no simultaneous communication between the parties involved. This approach has proven particularly effective during the recent COVID-19 pandemic, minimizing risks and improving clinical outcomes. In addition, it has proven to be a safe way to monitor clinical parameters, with the possibility of personalized and timely intervention for patients with chronic conditions, leading to improved patient condition and quality of life, while also helping to reduce costs for both the patient and the healthcare system. Asynchronous telemedicine and/or telerehabilitation activities, in which the patient and operator are not online at the same time, also enable patients living in remote areas with limited or unreliable connectivity to receive convenient, flexible, and accessible healthcare services.

DETAILED DESCRIPTION:
The project, considering the impact of robotic rehabilitation and asynchronous telerehabilitation on cognitive-motor interference, is highly innovative in terms of the integrated use of technology to improve the quality of life of frail people. Through the proposed therapeutic protocol, it will be possible to further customize the recommended rehabilitation treatments, both in outpatient and home settings, considering the characteristics of the patient and the evolution of the clinical picture. The use of telerehabilitation tools, used asynchronously, will allow greater access to care and widespread rehabilitation throughout the territory, including areas that are difficult to reach or from which patients and their caregivers have difficulty traveling.

The proposed technology, both in the home and outpatient settings, will be able to provide the patient with different types of real-time feedback (visual, auditory, tactile) to increase the level of interaction and involvement with the patient during rehabilitation treatment. In the outpatient setting, this feedback, combined with the constant presence of the physical therapist, will guide the patient during the exercise and various rehabilitation activities proposed. In the home setting, this feedback, combined with telephone monitoring by the healthcare professional, will ensure that the patient does not feel abandoned during the telerehabilitation treatment period, but receives care that is as similar as possible to that provided in an outpatient setting. The integration and synoptic interpretation of data collected with clinical and home technologies will enable better management of the care pathway, allowing for objective performance assessment and the subsequent delivery of personalized and specific treatments for each patient.

The main innovation of the project is the integration and combination of different robotic and technological products: the development of a rehabilitation pathway that ensures continuity between the clinic and the home will lead to the development of a new rehabilitation paradigm that is easily accessible to frail people.

Currently, the scientific literature offers a wide range of scientific articles on robotic rehabilitation and telerehabilitation, but there is still insufficient scientific evidence on the integrated use of outpatient robotic rehabilitation and home-based telerehabilitation, especially in frail individuals with chronic sensorimotor and/or cognitive disorders, particularly with regard to the impact on the simultaneous performance of motor and cognitive tasks. The results obtained from this project will fill the gap in the literature, allowing the dissemination of new knowledge and the development of a new rehabilitation paradigm.

With this in mind, the overall objective of the project will be to identify a new multi-perspective rehabilitation paradigm/pathway that can contribute to improving and maintaining residual cognitive and motor abilities in frail subjects in the chronic phase of the disease in the medium term. For this reason, a multicentre rehabilitation project will be developed that involves the use of innovative and integrated technological tools for both outpatient and asynchronous home rehabilitation.

The project will target frail individuals with chronic sensorimotor and/or cognitive disorders and will focus on the development of a rehabilitation paradigm to be integrated into the existing territorial ecosystem. As already mentioned, the aim of the project is to conduct a multicentre study focused on outpatient and home-based technological rehabilitation, with the main objective of identifying an innovative technological rehabilitation pathway aimed primarily at frail individuals with chronic sensorimotor and/or cognitive deficits and, in particular, at improving cognitive-motor interference, i.e., improving the ability to perform two tasks simultaneously, one cognitive and one motor. The reduction, understood as improvement, of cognitive-motor interference will have a positive impact on the quality and/or speed of execution of certain activities of daily living, indirectly influencing the quality of life of frail individuals, caregivers, and family members.

The specific objectives of the project will be, in line with Mission 1, to evaluate the effectiveness of the proposed rehabilitation paradigm in terms of improved clinical outcomes, patient satisfaction, treatment adherence, and trust and acceptance of the technology used. To achieve these specific objectives, a multicentre, randomized, single-blind, controlled clinical study will be designed to evaluate the clinical and economic feasibility of a technological rehabilitation treatment in outpatient and home settings in improving and/or maintaining certain specific functions, compared to conventional rehabilitation treatment (outpatient and home) in a group of frail subjects.

Patients will be recruited from the Post-Acute Rehabilitation Unit of the A. Gemelli IRCCS University Hospital in Rome and the Moderata Durant Polyclinic in Vibo Valentia who meet the inclusion criteria. Patients will be divided into two groups by randomization, as specified below. One group (G-Tec) will undergo outpatient technological rehabilitation treatment for 4 weeks, followed by 4 weeks of home-based technological rehabilitation treatment, and then 8 weeks of observation; the other group (G-Con) will undergo conventional outpatient rehabilitation treatment for 4 weeks, followed by 4 weeks of conventional home rehabilitation treatment, and then 8 weeks of observation. This project aims to implement a multicentre, randomized, controlled, single-blind, medical device clinical trial lasting 18 months.

All patients deemed eligible will be randomized into two groups (as described below): G-Tec patients will undergo 4 weeks of outpatient technological rehabilitation treatment (T0-T1) using the hunova® and Senso robots, followed by home-based technological rehabilitation treatment for another 4 weeks (T1-T2) using a tablet with cognitive exercises developed specifically for home-based cognitive treatment, followed by 8 weeks of observation (T2-T3); G-Con patients will undergo conventional outpatient rehabilitation treatment for 4 weeks (T0-T1), followed by conventional home-based rehabilitation treatment, mainly cognitive in nature, for another 4 weeks (T1-T2), and then 8 weeks of observation (T2-T3).

The rehabilitation protocol is specifically divided into 3 different phases. PHASE I. The first phase is outpatient rehabilitation (T0-T1): during this phase, all patients deemed eligible and randomized to G-Tec or G-Con will undergo outpatient rehabilitation treatment for 4 weeks, 45 minutes a day, 3 times a week. G-Tec patients will undergo rehabilitation treatment using robotic (hunova®, Movendo Technology Srl) and technological (Senso, THERA-Trainer) tools. G-Con patients, on the other hand, will undergo the same exercises as G-Tec patients, but these will be performed according to conventional rehabilitation activities. Patient satisfaction, adherence to treatment, and acceptance of the technology used (using TAM) will be assessed by an operator responsible for collecting this information. The sustainability of the treatment will be evaluated at the end of this phase in terms of clinical efficacy (through multi-perspective assessment), access to rehabilitation and technology, and economic sustainability of the treatment.

PHASE II. The second phase of the project is the home rehabilitation phase (T1-T2): G-Tec patients will undergo 4 weeks of asynchronous home telerehabilitation, 45 minutes a day, 3 times a week, using technological tools that can be used at home to carry out rehabilitation treatment aimed at improving, enhancing, or maintaining residual cognitive abilities. During this phase, G-Con patients will undergo home-based cognitive treatment equivalent to that offered to G-Tec patients, according to specific instructions provided by their doctor and physical therapist. Specifically, G-Tec patients will receive a tablet with the Rehability neuro software (Imaginary srl, Milan, Italy) containing cognitive exercises to be performed at home, while seated (asynchronously) and without supervision; the cognitive exercises will be preloaded by the operator onto the device, which will then be given to the patient. G-Con patients will receive a booklet of cognitive exercises to be performed at home, while seated. Rehability neuro is software classified as a Class I Medical Device, developed as a gaming tool for telerehabilitation. An internet connection will be required for the exercises to be delivered correctly, so patients will be provided with a device (commercial tablet) capable of using a WiFi connection (the tablets will not be equipped with 4G technology). Rehability neuro can be viewed on a tablet, with the patient performing the exercises in a seated position, or using the home kit connected to the TV. In this study, the Rehability Neuro software will be used in its tablet version, with the patient playing in a seated position, without using the home kit. The interface for clinical staff allows them to create a profile for each patient, recording the patient's data in a pseudo-anonymous form (only the ID and gender will be entered). Once the patient profile has been created, a rehabilitation plan can be associated with it, allowing structured exercises to be performed to stimulate cognitive functions such as attention, short-term memory, executive functions, visual processing, and response speed. After creating the game plan, it must be associated with a specific device, specifying the start and end dates of the plan (4 weeks) and the specific training days (3 days per week), as well as other information such as the order of the games (information such as calibration and fluidity will not be considered for the performance of activities on tablets and will therefore not be set). At the end of each game session, a report will be automatically generated, which will include information such as the actual execution of the session, the number of games completed, the cumulative score achieved, and information about the individual game (score, correct targets, incorrect targets). The tablet version of Rehability Neuro does not allow you to record parameters such as posture or physiological parameters, only data relating to the games played (number of games, score, etc.). Once the exercises have been associated with the device, each patient will be given a username (corresponding to the study ID) and password to access the game session through the application installed on the tablet. Using the tablet version of the software, it will not be possible to choose how to play (keyboard, mouse, Kinect, etc.) on the home page, but the patient will be redirected directly to the screen containing the games. During each game, the patient will receive visual and auditory feedback to highlight whether their actions are correct or not, helping them to understand their progress and correct themselves. At the end of each exercise, the final score for the exercise will be displayed. The Rehability neuro software will provide games such as: "Catch a mole," "Pedal bin," "Recycling," "Masterchef," "Moveat," "Breadbuster," "Guess the match," "Driving license," "Red dots," "Shapes and colors," "Fish and jellyfish," "Deep blue," "Rockets and meteorites," "Rockets and meteorites," "Rockets and meteorites," "Popping flowers," "Colored cans," "Magnetic maze," "Mad fridge," "Shopping bags," "Four seasons," "Find it," "Match it," "Solve it," and "Complete it." Each activity will be accompanied by an explanation in Italian of the exercises to be performed. The raw data from the exercises collected through the Rehability neuro software will only be available to operators at the end of the home gaming period, when the patient returns to the center to return the device (T2). At this stage, the effectiveness of the treatment will be assessed at T2 through a multi-perspective clinical and instrumental evaluation carried out by an expert operator. Patient satisfaction and acceptability of the technology will also be assessed at the end of the second phase by an operator responsible for collecting this information, including through the use of validated questionnaires (TAM). Adherence to treatment will be assessed in two ways: both through information collected by the operator, who will have weekly telephone contact with the enrolled patients, and through the collection of log data using the technology used at home (especially for G-Tec patients).

PHASE III. The third and final phase is the follow-up phase, which lasts 8 weeks (T2-T3): in this phase, patients enrolled in the study, whether allocated to G-Tec or G-Con, will not undergo rehabilitation treatment. The effectiveness of the treatment, understood in this phase as the maintenance of the improvements achieved in the first two phases, will be documented at the end of the follow-up period through a multi-perspective clinical and instrumental assessment carried out by an expert operator. For this phase, there is no assessment of adherence to rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 90 years;
* Presence of chronic sensorimotor and/or cognitive disabilities;
* Cognitive abilities that allow the patient to carry out simple orders and understand the physiotherapist's instructions [assessed using the Token Test (score ≥ 26.5)];
* Ability to walk independently or with minimal assistance;
* Ability to understand and sign the informed consent form.

Exclusion Criteria:

* Presence of systemic, neurological, or cardiac conditions that make walking risky or cause motor deficits;
* Oncological conditions, orthopedic or postural problems, presence of plantar ulcers;
* Partial or total amputation of segments of the foot.
* Inability to provide informed consent.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Dual-Task Cost (DTC) | Change from Baseline DTC at 8 weeks
  DTC refers to the deterioration in performance in one or both tasks when two tasks are performed simultaneously compared to when they are performed individually. This cognitive cost manifests itself as a reduction in speed, accuracy or quality in task performance, and can be measured by comparing individual performance with that achieved in "dual task" mode. Specifically, DTC is calculated as the difference between the displacement of the centre of pressure during a cognitive task and the displacement of the centre of pressure during a single-task activity with eyes open, divided by the displacement of the centre of pressure during a single-task activity with eyes open.
  Higher DTC values correspond to a deterioration in performance.

SECONDARY OUTCOMES:
Hand Grip Strength Test (HSGT) | Change from Baseline HGST at 8 weeks
  HGST is a test performed with a dynamometer, which goes to assess muscle strength (in kilograms). Starting with the elbow flexed to 90° the patient must squeeze the dynamometer as hard as they can at one time. Three repeated measurements are taken on each side 20 seconds apart. The average of the three assessments is used as the final value.
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 8 weeks
  SPPB is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). Three domains, which include balance, usual or self-selected gait speed, and lower limb strength, are assessed by a three-stage balance test (feet side-by-side, semitandem, and tandem positions), a 3-m or 4-m gait speed test (time spent to walk the course), and a repetitive chair stand test (five times chair sit-to-stand test), respectively. A 0- to 12-point scale is used to score the sum of the three assessments with higher point values corresponding with greater levels of physical function and lower disability, whereas lower point values correspond with lower levels of physical function and higher disability, respectively.
Timed Up and Go Test (TUG) | Change from Baseline TUG at 8 weeks
  The Timed Up and Go test (TUG) measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down. The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 is severely abnormal) according to the observer's perception of the patient's risk of falling. The timed part of the test records the mean time (in seconds) from initial getting up to re-seating. Patients are compared with the mean time of adults in their age group, 60 to 69, 70 to 79, and 80 to 99 years of age.
Six-minute walk test (6MWT) | Change from Baseline 6MWT at 8 weeks
  The 6MWT is a sub-maximal exercise test used to assess walking endurance and aerobic capacity. Participants will walk around the perimeter of a set circuit for a total of six minutes. The score of the test is the distance a patient walks in 6 minutes (measured in meters and can round to the nearest decimal point). Distance (in meters) covered in six minutes is calculated by multiplying the number of total laps by 12 meters and adding the distance of the partial lap completed at the time the test ended.
Timed-25 Foot Walk (T25FW) | Change from Baseline T25FW at 8 weeks
  The T25FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Silver Index (SI) | Change from Baseline SI at 8 weeks
  The SI is an objective test to identify the risk of falling, which is carried out using the Hunova robotic platform. It consists of seven domains: (i) static balance (ii) dynamic balance (iii) reactive balance (iv) sensory integration (v) stability limits (vi) sitting-to-standing position (vii) gait speed. At the end of the evaluation you get a percentage that indicates the risk of falling: higher percentages correspond to a higher risk of falling.
Trial Making Test (TMT) | Change from Baseline TMT at 8 weeks
  The Trail Making Test (TMT) measures flexibility of thinking on a visual-motor sequencing task. It consists of two parts, A and B, where 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment. Trail A: Average 29 seconds, Deficient > 78 seconds, Rule of Thumb Most in 90 seconds Trail B: Average 75 seconds, Deficient > 273 seconds, Rule of Thumb Most in 3 minutes.
Symbol Digit Modalities Test (SDMT) | Change from Baseline SDMT at 8 weeks
  The Symbol Digit Modalities Test (SDMT) is a test that assesses information processing speed and consists of a series of nine printed symbols to which nine numbers correspond. After a 'training' phase, patients are asked to match as many symbols as possible to the corresponding number in just 90 seconds. As the test persons can give written or oral answers, the test is suitable for people with motor disabilities or speech disorders. The score is calculated by adding up the number of correct substitutions in the 90-second interval (maximum = 110). Interpretation results from normalising the categories of gender, age and education.
Stroop Colour Word Test (SCWT) | Change from Baseline SCWT at 8 weeks
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. The subject is asked to read the words in the first task, to name colors in the second and third tasks. It is necessary to mark both any mistakes made but also the time spent on each task. The cut-off for the error interference effect is 4.24, while the cut-off for the time interference effect is 36.92.
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 8 weeks
  The Modified Fatigue Impact Scale (MFIS) is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items. The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument. The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.
EuroQoL- 5D (EQ-5D) | Change from Baseline EQ-5D at 8 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline HADS at 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a tool used to check for symptoms of anxiety and depression, especially in hospital patients. It has 14 questions, 7 for anxiety and 7 for depression. Each question is scored from 1 to 4.
Pittsburgh Sleep Quality Index (PSQI) | Change from Baseline PSQI at 8 weeks
  The PSQI is a sleep quality assessment scale that considers the last month; it consists of 19 items that must be assessed by the subject themselves and another 5 that must be completed by their bed or room partner (which are not included in the total score, but serve only as clinical information).
  In calculating the PSQI score, seven composite scores are derived (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of hypnotic medications, daytime disturbances), each with a score from 0 (no difficulty) to 3 (severe difficulty). The scores for the 7 domains are added together to produce an overall score (from 0 to 21). Higher scores indicate poorer sleep quality.
Bioimpedance analysis (BIA) | Change from Baseline BIA at 8 weeks
  BIA measures phase angle (PhA), which is related to cellular health and muscle quality. Lower PhA values have typically been observed in individuals with serious medical conditions and have been linked to poorer outcomes; conversely, higher PhA values are indicative of better overall health, strength, and muscle function.
SARC-F | Change from Baseline SARC-F at 8 weeks
  The SARC-F is a simple screening tool used to identify individuals at risk of sarcopenia. It consists of 5 questions assessing strength, assistance with walking, rising from a chair, climbing stairs, and falls. Each item is scored from 0 to 2, with a total score ranging from 0 to 10. A score of 4 or higher suggests a risk of sarcopenia and the need for further assessment.
Mini Nutritional Assessment- short Form (MNA-SF) | Change from Baseline MNA-SF at 8 weeks
  The Mini Nutritional Assessment - Short Form (MNA-SF) is a screening tool used to quickly evaluate the risk of malnutrition in older adults. It consists of 6 questions covering aspects such as weight loss, appetite, mobility, psychological stress, and body mass index (BMI) or calf circumference. Scores range from 0 to 14, with 12-14 indicating normal nutrition, 8-11 at risk of malnutrition, and 0-7 indicating malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy
  - Poliambulatorio Moderata Durant, Vibo Valentia, VV